CLINICAL TRIAL: NCT04660344
Title: A Phase III, Double-blind, Multicenter, Randomized Study of Atezolizumab (Anti-PDL1 Antibody) Versus Placebo as Adjuvant Therapy in Patients With High-risk Muscle-invasive Bladder Cancer Who Are ctDNA Positive Following Cystectomy
Brief Title: A Study of Atezolizumab Versus Placebo as Adjuvant Therapy in Participants With High-risk Muscle-invasive Bladder Cancer (MIBC) Who Are ctDNA Positive Following Cystectomy
Acronym: IMvigor011
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO42843; 2020-004418-36 (EudraCT Number); 2022-502705-15-00 (EU CTIS Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Muscle-invasive Bladder Cancer
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Atezolizumab (Experimental): Atezolizumab will be administered intravenously (IV) at a dose of 1680 milligrams (mg) on Day 1 of each 28-day cycle for 12 cycles or up to 1 year (whichever occurs first). Atezolizumab will be discontinued in the event of disease recurrence, unacceptable toxicity, withdrawal of consent, or study termination by the Sponsor.
  Interventions: Drug: Atezolizumab; Device: Signatera
- Arm B: Placebo (Placebo Comparator): Placebo will be administered IV on Day 1 of each 28-day cycle. Placebo will be discontinued in the event of disease recurrence, unacceptable toxicity, withdrawal of consent, or study termination by the Sponsor.
  Interventions: Other: Placebo; Device: Signatera
- Arm C: Surveillance Follow-Up (Experimental): Participants who remain ctDNA negative at 12 months from the date of cystectomy will not be randomized to treatment and will enter follow-up.
  Interventions: Device: Signatera

INTERVENTIONS:
Drug: Atezolizumab — ctDNA positive participants will receive 1680 mg IV, every 4 weeks (Q4W) on Day 1 of each 28-day cycle.
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab
Other: Placebo — ctDNA positive participants will receive placebo IV, Q4W on Day 1 of each 28-day cycle
  Arms: Arm B: Placebo
Device: Signatera — Signatera will be used to evaluate whether ctDNA is detected during serial monitoring of peripheral blood samples for participants enrolled in surveillance. Participants with a ctDNA positive result will be screened for inclusion in the treatment phase. Participants who remain ctDNA negative at 12 months from the date of cystectomy will not be randomized to treatment and will enter follow-up.

SUMMARY:
This is a global Phase III, randomized, placebo-controlled, double-blind study designed to evaluate the efficacy and safety of adjuvant treatment with atezolizumab compared with placebo in participants with MIBC who are circulating tumour deoxyribonucleic acid (ctDNA) positive and are at high risk for recurrence following cystectomy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Surveillance Phase:

* Histologically confirmed MIUC (also termed transitional cell carcinoma [TCC]) of the bladder
* Tumor, nodes, and metastases (TNM) classification (based on American Joint Committee on Cancer [AJCC] Cancer Staging Manual, 8th Edition; Amin et al. 2016) at pathological examination of surgical resection specimen as follows: For participants treated with prior neoadjuvant chemotherapy (NAC): tumor stage of ypT2-4a or ypN+ and M0. For participants who have not received prior NAC: tumor stage of pT2-4a or pN+ and M0
* Surgical resection of MIUC of the bladder
* Participants who have not received prior platinum-based NAC must be ineligible for cisplatin-based adjuvant chemotherapy, have refused it, or will not receive it based on physician's decision
* ctDNA assay developed based on tumor tissue specimen and matched normal DNA from blood
* Tumor programmed death ligand (PD-L1) expression per immunohistochemistry (IHC) that is evaluable by central testing of a representative tumor tissue specimen
* Absence of residual disease and absence of metastasis, as confirmed by a negative baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan of the pelvis, abdomen, and chest no more than 4 weeks prior to enrollment
* Full recovery from cystectomy and enrollment within 24 weeks following cystectomy. Minimum of 6 weeks must have elapsed from surgery

Additional Inclusion Criteria for the Treatment Phase:

* Blood for plasma ctDNA sample evaluated to be ctDNA positive, defined as the presence of two or more mutations out of the 16 mutations identified based on participant' whole exome sequencing (WES) evaluable (ctDNA assay designability) report
* Absence of residual disease and absence of metastasis, as confirmed by a negative baseline CT or MRI scan of the pelvis, abdomen, and chest no more than 28 days prior to randomization, as assessed by the investigator and Independent Review Facility
* Eastern cooperative oncology group (ECOG) performance status of ≤ 2
* Life expectancy ≥12 weeks
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs

Exclusion Criteria:

General Medical Exclusion Criteria for the Surveillance Phase:

* Known PD-L1 IHC result for adjuvant therapy. The decision for the adjuvant therapy should not be based on the PD-L1 IHC result
* Pregnancy or breastfeeding
* Positive test for human immunodeficiency virus (HIV), with the following exception: Participants with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy, have a cluster of differentiation 4 (CD4) count ≥ 200 per microliter (/µL), and have an undetectable viral load
* Participants with active hepatitis B virus (HBV) or hepatitis C virus (HCV). Participants with past HBV infection or resolved HBV infection are eligible. A negative HBV deoxyribonucleic acid (DNA) test must be obtained in these participants prior to enrollment. Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Active tuberculosis (TB) confirmed by a test performed within 3 months prior to treatment initiation
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease. Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study. Participants with controlled type I diabetes mellitus (T1DM) on a stable dose of insulin regimen may be eligible for this study
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction (MI) within the previous 3 months, unstable arrhythmias, or unstable angina

Cancer-Specific Exclusion Criteria for the Surveillance Phase:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to study enrollment
* Adjuvant chemotherapy or radiation therapy for UC following cystectomy
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or 5 half-lives of the drug, whichever is longer, prior to enrollment
* Malignancies other than UC within 5 years prior to study enrollment

Additional Exclusion Criteria for the Treatment Phase:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to randomization to the treatment phase. Hormone-replacement therapy or oral contraceptives are allowed
* Adjuvant chemotherapy or radiation therapy for UC following cystectomy
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or 5 half-lives of the drug, whichever is longer, prior to randomization to the treatment phase
* Positive test for HIV, with the following exception: Participants with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy, have a CD4 count ≥200/μL, and have an undetectable viral load
* Participants with active HBV or HCV
* Active tuberculosis confirmed by a test performed within 3 months prior to treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-09-13 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed (INV) - Disease-free Survival (DFS) | Randomization up to first occurrence of DFS event (up to approximately 40 months)
  INV-DFS, defined as the time from randomization to the first occurrence of a DFS event, defined as any of the following:
  * Local (pelvic) recurrence of urothelial carcinoma (UC) (including soft tissue and regional lymph nodes);
  * Urinary tract recurrence of UC (including all pathological stages and grades);
  * Distant metastasis of UC;
  * Death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Randomization up to death from any cause (up to approximately 10 years)
  OS, defined as the time from randomization to death from any cause.
Independent Review Facility (IRF)-assessed DFS | Randomization up to first occurrence of DFS event (up to approximately 40 months)
INV Disease-specific Survival (DSS) | Randomization to death from UC (up to approximately 10 years)
  INV-DSS, defined as the time from randomization to death from UC per investigator assessment of cause of death.
INV Distant Metastasis-free Survival (DMFS) | Randomization to diagnosis of distant metastases or death from any cause (up to approximately 10 years)
  INV-DMFS, defined as the time from randomization to the diagnosis of distant (i.e., non-locoregional) metastases or death from any cause.
Time to Confirmed Deterioration of Function and Health-related Quality of Life (HRQoL) | Randomization to participant's first score decrease of ≥ 10 points from baseline on EORTC QLQ-C30 physical function scale, role function scale, and the GHS/QoL Scale (up to approximately 10 years)
  Time to confirmed deterioration of function and HRQoL, defined as the time from randomization to the date of a participant's first score decrease of ≥ 10 points from baseline on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) physical function scale, role function scale, and the global health status (GHS)/QoL scale (separately), held for at least two consecutive time points or followed by death.
ctDNA Clearance | Baseline, Cycle 3 Day 1 or Cycle 5 Day 1 (each cycle is 28 days)
  ctDNA clearance, defined as the proportion of participants who are ctDNA positive at baseline and ctDNA negative at Cycle 3, Day 1 or Cycle 5, Day 1.
Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 10 years
Serum Concentration of Atezolizumab | At pre-defined intervals from first administration of study drug (up to approximately 10 years)
Incidence of Anti-Drug Antibodies (ADAs) to Atezolizumab | Baseline up to approximately 10 years
  Incidence of ADAs to atezolizumab after initiation of study treatment (postbaseline incidence).
Prevalence of ADAs to Atezolizumab | Baseline
  Prevalence of ADAs to atezolizumab at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (161):
- United States (7):
  - UCLA Department of Medicine, Santa Monica, California
  - Rocky Mountain Cancer Center - Denver, Littleton, Colorado
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - Optum Health Care, Las Vegas, Nevada
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - AHN Cancer Institute ? Allegheny General Hospital, Pittsburgh, Pennsylvania
- Argentina (2):
  - Centro Medico Austral, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
- Belgium (3):
  - AZ KLINA, Brasschaat
  - UZ Gent, Ghent
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (10):
  - Oncocentro Serviços Medicos E Hospitalares Ltda, Fortaleza, Ceará
  - CETUS Hospital Dia Oncologia, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - *X*Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- China (15):
  - Friendship Hospital, Capital Medical University, Beijing
  - the First Hospital of Jilin University, Changchun
  - Hu Nan Provincial Cancer Hospital, Changsha
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - Yantai Yu Huangding Hospital, Yantai
- Colombia (3):
  - Clinica del Country, Bogotá
  - Instituto Cancerología Medellin, Medellín
  - Oncomedica S.A., Montería
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
  - Fakultni Thomayerova nemocnice, Praha 4 - Krc
- France (11):
  - ICO Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hopital Saint Andre, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Centre D'Oncologie de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Institut Mutualiste Montsouris, Paris
  - Hopital Foch, Suresnes
  - Institut Claudius Régaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Urologie, Halle
  - Universitätsklinikum der Ruhr-Universität Bochum, Marien-Hospital Herne, Urologische Klinik, Herne
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Greece (5):
  - Attikon University General Hospital, Ahens
  - Alexandras General Hospital of Athens, Athens
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras Medical Oncology, Pátrai
  - Theageneio Hospital, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Ireland (2):
  - Cork Uni Hospital, Cork
  - Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital, Dublin
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (13):
  - Azienda Ospedaliera di Rilievo Nazionale "Antonio Cardarelli", Day Hospital Oncologico, Napoli, Campania
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale, Napoli, Campania
  - AZ.Osp S. Orsola ? Malpighi-Reparto di Oncologia Medica, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Policlinico Universitario "Agostino Gemelli", Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - A.O. Universitaria S. Luigi Gonzaga, Orbassano, Piedmont
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato, Arezzo, Tuscany
  - Azienda Ospedaliera Santa Maria di Terni, Terni, Umbria
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Japan (23):
  - Nagoya University Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Shikoku Cancer Center, Ehime
  - Kyushu University Hospital, Fukuoka
  - Fukuyama City Hospital, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - St. Marianna University Hospital, Kanagawa
  - Yokosuka Kyosai Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Nagano Municipal Hospital, Nagano
  - Iwate Medical University Hospital, Numakunai
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Tokushima University Hospital, Tokushima
  - National Cancer Center Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Toyama University Hospital, Toyama
- CUAN Hospital, San Pedro Garza García, Nuevo León, Mexico
- Poland (4):
  - PRATIA MCM Kraków, Krakow
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu, Późna
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroc?aw
- Russia (5):
  - St-Petersburg Regional Oncology Dispensary, Kuzmolovo, Leningrad
  - Privolzhsk Regional Medical Center, Nizhny Novgorod, Niznij Novgorod
  - FSI Russian Centre of Radiology and Surgical Technologies, Saint Petersburg, Sankt-Peterburg
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Murmansk Regional Clinical Hospital named after P.A. Bayandin, Murmansk
- National Cancer Centre, Singapore, Singapore
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (14):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Turkey (Türkiye) (9):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Ankara University Faculty of Medicine Cebeci Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul
  - Medeniyet University Goztepe Training and Research Hospital., Istanbul
  - Medikal Park Izmir Hospital, Kar??yaka
  - Medikal Park Samsun, Samsun
- Ukraine (5):
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval Department of Urology #4, Kharkiv, Kharkiv Governorate
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC SI Dnipropetrovsk MA of MOHU Ch of Oncology and MR, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center, Kyiv
- United Kingdom (11):
  - Addenbrookes Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Barts Hospital, London
  - University College London NHS Foundation Trust, London
  - Royal Marsden Hospital - London, London
  - Charing Cross Hospital, London
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Weston Park Hospital, Sheffield
  - Southampton University Hospitals NHS Trust, Southampton
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Powles T, Kann AG, Castellano D, Gross-Goupil M, Nishiyama H, Bracarda S, Bjerggaard Jensen J, Makaroff L, Jiang S, Ku JH, Park SH, Reig Torras O, Ye D, Maruzzo M, Necchi A, Morales-Barrera R, Giunta EF, Lee JL, Tortora G, Urun Y, Dolowy L, Erdem D, Pinto A, Grando F, Zou W, Assaf ZJ, Vuky J, Degaonkar V, Steinberg EE, Bellmunt J, Gschwend JE; IMvigor011 Investigators. ctDNA-Guided Adjuvant Atezolizumab in Muscle-Invasive Bladder Cancer. N Engl J Med. 2025 Dec 18;393(24):2395-2408. doi: 10.1056/NEJMoa2511885. Epub 2025 Oct 20. PMID 41124204
- [Derived] Jackson-Spence F, Toms C, O'Mahony LF, Choy J, Flanders L, Szabados B, Powles T. IMvigor011: a study of adjuvant atezolizumab in patients with high-risk MIBC who are ctDNA+ post-surgery. Future Oncol. 2023 Mar;19(7):509-515. doi: 10.2217/fon-2022-0868. Epub 2023 Apr 21. PMID 37082935